CLINICAL TRIAL: NCT00910741
Title: Phase I/II Study of the Combination Therapy With NC-6004 and Gemcitabine in Patients With Locally Advanced or Metastatic Pancreatic Cancer in Asian Countries
Brief Title: NC-6004(Nanoplatin) and Gemcitabine to Treat Pancreatic Cancer in Asia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanoCarrier Co., Ltd. (Industry)
Collaborators: Orient Europharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-6004-002
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Locally Advanced and Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — demplatin pegraglumer; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nanoplatin (Experimental): Nanoplatin (NC-6004) had to be administered once every 3 weeks, on Day 1, Day 22 and Day 43 etc.
  Gemcitabine had to be administered to every patient 2 times on Day 1 and Day 8 every 3 weeks after the infusion of Nanoplatin (NC-6004).
  Interventions: Drug: Nanoplatin (NC-6004) and Gemcitabine

INTERVENTIONS:
Drug: Nanoplatin (NC-6004) and Gemcitabine

SUMMARY:
The purpose of this study is to determine the recommended dose of NC-6004 according to the dose-limiting toxicity (DLT) in combination with Gemcitabine, and to assess the efficacy, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chemo-naive, advanced pancreatic cancer
* Nonresectable, histologically or cytologically confirmed, locally advanced or metastatic pancreatic cancer

Exclusion Criteria:

* Pulmonary fibrosis or interstitial pneumonia
* Marked pleural effusion or ascites above Grade 2
* Severe drug hypersensitivity
* Metastasis to the central nervous system and brain

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT and Response rate | DLT is evaluated for 3 weeks o the treatment, Response rate is evaluated at 7,13,19 and 25weeks of the treatment

SECONDARY OUTCOMES:
Overall survival | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (5):
- National Cancer Centre Singapore, Singapore, Singapore
- Taiwan (4):
  - Natinal Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veteran General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Background] Uchino H, Matsumura Y, Negishi T, Koizumi F, Hayashi T, Honda T, Nishiyama N, Kataoka K, Naito S, Kakizoe T. Cisplatin-incorporating polymeric micelles (NC-6004) can reduce nephrotoxicity and neurotoxicity of cisplatin in rats. Br J Cancer. 2005 Sep 19;93(6):678-87. doi: 10.1038/sj.bjc.6602772. PMID 16222314